CLINICAL TRIAL: NCT03256929
Title: Personalized Diet-driven Microbiota Alterations as a Tool for Improving Mood Status in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Hai College (Other)
Collaborators: Shamir Research Institute (Unknown); Clalit Health Services (Other); Migal, Galilee Technology Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHAMIRMB
Record Dates: First submitted 2017-08-12; First posted 2017-08-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: Personalized Diet; Microbiota; Depression; Elderly; Gut flora
MeSH Terms: conditions — Depression | interventions — Health

STUDY DESIGN:
Intervention Model Description: The first stage will be mapping all of the aged population of the research area, who will be interviewed (after receiving their consent) in order to determine those who are depressed. 200 depressed and pre-depression individuals (according to the GDS) will be chosen, and divided randomly into two groups- one will undergo the diet- driven microbiota adjustment personalized-intervention (nutrition advisory), and the other will get general information on nutrition and health .
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- depression participants - intervention (Experimental): personalized diet intervention based on microbiota analysis and health status
  Interventions: Behavioral: Personalized Diet-driven microbiota
- depression participants - control (Experimental): General information on nutrition and health
  Interventions: Behavioral: General information on nutrition and health
- pre-depression participants - control (Experimental): General information on nutrition and health for pre-depression participants
  Interventions: Behavioral: General information on nutrition and health
- pre-depression participants - intervention (Experimental): personalized diet intervention based on microbiota analysis and health status for pre-depression participants
  Interventions: Behavioral: Personalized Diet-driven microbiota

INTERVENTIONS:
Behavioral: Personalized Diet-driven microbiota — Based on the results of the individual microbiota profile, the investigators will formulate a specific diet aiming to enrich the distinct microbiota with organisms correlated to better mental health. The dietitian will visit each participant twice a month.
  Arms: depression participants - intervention; pre-depression participants - intervention
Behavioral: General information on nutrition and health — General information on nutrition and health. The dietitian will visit each participant twice a month.
  Arms: depression participants - control; pre-depression participants - control

SUMMARY:
The propose of the study is a multi-disciplinary project connecting nutritional and health sciences with social and behavioral sciences, and aimed at understanding the microbiota changes related to the third age and their effects on mood and mental health. The research aims are primarily practical: They will explore the influence of the gut flora on depression, which could help us to recommend diets that might reduce the risk of developing depression. The novelty of this proposal is in the design of personalized diet-driven microbiota alterations and health status to modulate depression in elderly. For the first time the improvement of mental health in the elderly will be studied through a nutritional and food habits approach based on microbiota changes upon ageing.

DETAILED DESCRIPTION:
Depressive symptoms are highly prevalent in older populations, is one of the most serious public health problems faced by modern societies. The problems caused by depression, such as functional impairments, lead to decreased quality of life, poor recovery from illnesses and increased mortality in the elderly. Researchers have found that there are many possible connections between personal or physical variables and the risk of developing depression; it can be caused by sociodemographic factors, or cognitive and functional impairment, nutritional status is also related to development of depression.

Recent studies have suggested that depressive symptoms are more prevalent in individuals with impaired nutritional status. The intestinal microbial population (microbiota), known influenced by several factors including nutrition, age, and stress.

The microbiota is essential to human health, changes in composition microbiota play a role in metabolic, nutritional, physiological and immunological processes in the human body, recently reported also behavioral changes associated with anxiety and depression. The aging process is characterized by a decrease intestinal transit time, as a result of dental problems, decrease in saliva activity, and efficiency of digestion and absorption leading to changes in the microbiota composition, which causes an increase in sensitivity to the development of chronic and inflammatory diseases. Although other factors undoubtedly contribute to mental health decline in the elderly, the association of the intestinal microbiota of older people with inflammation, the clear association between diet and microbiota and the recent report on the correlation between changes in microbiota and depression have led us to hypothesize that diet can shape microbiota, which then affect mood status in older people and decreased depressive symptoms.

The purpose of the study is to examine the effect of a custom diet based on the composition of the intestinal bacterial population (compared with a diet for a healthy lifestyle that is not based on a microbiotic profile), on moods and depression among the elderly.

Before and after the intervention, several tests will be carried out, using stool sample for microbiota analysis, salivary cortisol measurement and clinical information (GDS, life style habits, CEBQ, FFQ), These measures will indicate participants' clinical, nutritional and mental situation before and after in order to probe the diet intervention impact on microbiota and its correlation to mental health.

The infrastructure of this research includes several aspects - mood, health and nutrition status that are main parameters in life quality of the third age, and the research is based on the complementary cooperation of social and behavior sciences and nutrition and life sciences experts.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged 60 - 80, from northeastern Israel, Jewish, Druze and Arab populations, will be recruited. Only healthy, independent people who agreed to take part in the study and show depressive symptoms according to the Geriatrics Depression Scale.

Exclusion Criteria:

* Elderly people with depression who are drug-treated or elderly who are nursing his/her partner, and who are treated with antibiotics at least 4 weeks before taking fecal samples.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Mental health status - Depression | 1 year
  Depression will be assessed using the Geriatric Depression Scale (GDS). changes in test score

SECONDARY OUTCOMES:
Microbiota profile | 1 year
  Microbiota composition will be characterized from feces. The stool specimens will be collected and immediately put in buffer and stored at -20ºC for analysis and then will be kept at -80ºC in a locked freezer. The very low temperature is of significance to avoid variability in the stool bacterial composition and to preserve bacterial DNA in fecal samples. Total microbial DNA will be extracted using the PowerSoil DNA extraction kit (MoBio) and then submitted to 16S rRNA gene amplicon sequencing using paired end Illumina technology.
Salivary Cortisol | 1 year
  Salivary Cortisol Measurement - The sampling procedure is simple and non-invasive. The saliva sample will be collected by using the Salivettes and freezed as is. On the day of the assay, Salivette™ samples can be thawed and then centrifuged at low speed to separate the saliva sample from the gauze. The cortisol in saliva is remarkably stable and will be measured by the salivary cortisol kit.
life style habits | 1 year
  The life style habits questionnaire is based on MABAT ZAHAV, National Health and Nutrition Survey (Aged 60 and over) 2005-2006, Ministry of Health, Israel and includes demographic details, questions on health status, dental health, functional, cognitive and emotional states, use of medications and nutrition supplements, alcohol consumption, physical activity, smoking habits, eating and dieting patterns, nutritional knowledge and attitudes.
Nutritional data collection - Food Frequency Questionnaire - FFQ | 1 year
  Habitual dietary intake information that will be assessed using the Food Frequency Questionnaire (FFQ)
Eating Behavior Questionnaire - CEBQ | 1 year
  Appetite, gastrointestinal problems, and chewing and swallowing problems will be assessed using the Composite Eating Behavior Questionnaire (CEBQ)

OTHER OUTCOMES:
Anthropometric measure 1 | 1 year
  Measurements of body weight in kilograms
Anthropometric measure 2 | 1 year
  Change in body fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Ofran, M.D, MPH, Principal Investigator — Clalit Health Services; Snait Tamir, Prof., Principal Investigator — Migal, Galilee Technology Center; Shmuel Shamai, Prof., Principal Investigator — Shamir Research Institute; Adi Vitman- Schorr, Ph.D, Principal Investigator — Shamir Research Institute; Karen Jackson, Ph.D, Principal Investigator — Migal, Galilee Technology Center
Locations (1):
- Shamir Research Institute, Qatzrin, Israel, Israel

IPD SHARING:
Plan to Share IPD: No